CLINICAL TRIAL: NCT05172388
Title: Cardiopulmonary Health Effects of Indoor Air Purification and Other Indoor Environmental Conditions Among Young Healthy Adults in Beijing, China
Brief Title: Indoor Air Filtration and Young Adults Health Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, Furong Deng, MD & PhD, Professor, Deputy Director Department of Occupational & Environmental Health Sciences, Peking University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: IRB00001052-21109
Record Dates: First submitted 2021-11-30; First posted 2021-12-29 (Actual); Last update posted 2022-10-13 (Actual); Status verified 2022-10

CONDITIONS: Cardiopulmonary Diseases
MeSH Terms: conditions — Pulmonary Heart Disease | interventions — Air Filters

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Real purification (Active Comparator): Air purifier turned on.
  Interventions: Other: Air purifier
- Sham purification (Sham Comparator): Air purifier turned off.
  Interventions: Other: Air purifier

INTERVENTIONS:
Other: Air purifier — Real purification and sham purification would be conducted in the dormintory rooms (about 25 in total) of the study subjects for 4 days, following a randomized crossover design, which means a real air purifier and a sham purifier would be placed in the same dormintory room with a wash-out interval (15 days).

SUMMARY:
This study aims to explore the cardiopulmonary health effects of indoor air purification and other indoor environmental conditions among young healthy college students in Beijing, China.

DETAILED DESCRIPTION:
The present randomized, double-blind crossover study was conducted to investigate the cardiopulmonary health effects of air purification among 81 young healthy college students in Beijing, China. Real or sham purification was performed in the dormitories for 4 days, following a 15-day wash-out period in the intervals. During the study periods, the investigators collected indoor exposure levels of size-fractionated particulate matter (PM), black carbon (BC), noise, ozone, nitrogen dioxide, carbon dioxide, volatile organic compounds, temperature, relative humidity, illumination, and microorganism. Biological specimens (i.e., morning urine, fasting venous blood, exhaled breath condensate, and nasal mucus) were also collected and examined. Some important individual factors including demographical information (age, sex, height, weight, etc.), physical activity, sleep condition, mood and cognition, and food intake were also gathered using questionaire or anthropometric measurements, in order to control for the potential confounding effects. For further data analyses, air pollutants, noise, and other exposures would be controlled as confounders when addressing the health effects associated with air purification, and would also be used to explore their effects on cardiopulmonary health. The interaction effects of air pollutants, noise, and other exposures on cardiopulmonary health would also be explored.

ELIGIBILITY:
Inclusion Criteria:

* Living in Beijing for more than one consecutive years;
* College students between 18-28 years;

Exclusion Criteria:

* Current or past smokers;
* Body mass index (BMI) over 28.0 kg/m2.
* Alcohol addict;
* Having thoracic surgery history;
* History of diagnosed chronic disease;
* Hepatitis B / hepatitis C virus patient / carrier;
* Unwilling or unable to provide informed consent or cooperate with all research related procedures.

Ages: 18 Years to 28 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 81 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Changes in heart rate variability | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Including the standard deviation of all normal-to-normal R-R intervals (SDNN) in millisecond, standard deviation of sequential five-minute R-R interval means (SDANN) in millisecond, root-mean-square difference of successive normal R-R intervals (rMSSD) in millisecond, low frequency (LF) in squared millisecond, and high frequency (HF) in squared millisecond.
Changes in blood pressure | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Including the systolic blood pressure (SBP) in mmHg, diastolic blood pressure (DBP) in mmHg, and pulse pressure (PP) in mmHg.
Changes in pulmonary function | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Including forced expiratory volume in 1 s (FEV1) in liter, forced vital capacity (FVC) in liter, forced expiratory volume in 1 s (FEV1) / forced vital capacity (FVC) ratio, and peak expiratory flow (PEF) in liter per second.

SECONDARY OUTCOMES:
Changes in levels of airway inflammation | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Respiratory inflammation Fractional exhaled nitric oxide (FeNO) test would be conducted.
Changes in levels of C-reactive protein (CRP) | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Examining the C-reactive protein (CRP) in blood sample to characterize the levels of inflammation.
Changes in levels of 8-hydroxydeoxyguanosine (8-OHdG) | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Examining the 8-hydroxydeoxyguanosine (8-OHdG) in urine sample to characterize the levels of oxidative stress.
Changes in levels of sleep-related parameters | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Including time in bed in minute, total sleep time and sleep stage time in minute. The time in bed and total sleep time would be calculated to sleep efficiency in percentage.
Changes in levels of sleep-breathing parameters | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Including blood oxygen saturation in percentage and heart rate in bpm.
Changes in levels of cognitive function | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Including short-term memory and delayed memory in unit measured by the standard Stroop Test, as well as executive function in unit measured by the Harmonized Cognitive Assessment Protocol.
Changes in levels of cognitive function-related biomarkers | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Including serum brain derived nerve factor (BDNF) in ng/mL, S100B protein in ng/mL, and neuron-specific-enolase (NSE) in ng/mL.
Changes in levels of blood cell parameters | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Including white blood cells in unit, red blood cells in unit, and platelets in unit measured by blood routine examination.
Changes in levels of systematic inflammation and oxidative stress indicators | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Including interleukin-6 (IL-6) in unit, IL-8 in unit, IL-10 in unit, IL-13 in unit, IL-5 in unit, IL-1β in unit, IL-17A in unit, IL-12p70 in unit, tumor necrosis factor-α (TNF-α) in unit, interferon-γ (IFN-γ) in unit, monocyte chemoattratctant protein-1 (MCP-1) in unit, angiotensin II (Ang-II) in unit, superoxide dismutase (SOD) in unit, glutathione (GSH) in unit, nitric oxide levels (NOX) in unit.
Changes in levels of glucose metabolites in serum | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Serum samples were collected for targetted glucose metabolomics analysis using the gas chromatography and mass spectrometry (GC-MS).
Changes in levels of neurotransmitter metabolites in serum | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Serum samples were collected for targetted neurotransmitter metabolomics analysis using the gas chromatography and mass spectrometry (GC-MS).
Changes in levels of microbiomics in nasal mucus | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Nasal mucus samples were collected for microbiomics analysis to examine the microbial community abundance (α-diversity).
Changes in levels of microbiomics in EBC | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  EBC samples were collected for microbiomics analysis to examine the microbial community abundance (α-diversity).
Changes in levels of pituitary-related hormones | Baseline and after the completion of intervention period (a 4-day real purifier intervention or a 4-day sham purifier intervention)
  Including serum levels of cortisol, adreno-cortico-tropic-hormone (ACTH), and thyroid stimulating hormone (TSH).

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University, Beijing, China